CLINICAL TRIAL: NCT02917967
Title: A Pilot Study of the Effect of Botulinum Toxin Type a (Dysport®, Abobotulinum Toxin A) Injection on Changes in Musculotendinous Length and Dynamics of Hamstring Muscles During Gait in Children With Spastic Cerebral Palsy Walking With Excessive Knee Flexion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0265
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTX injection group (Experimental): Botulinum toxin injection group
  Interventions: Drug: Botulinum toxin injection

INTERVENTIONS:
Drug: Botulinum toxin injection — 1. BoNT-A will be injected into two hamstring and/or gastrocnemius muscles under the guidance of ultrasonography or electrical stimulation.
  2. Maximal total dose and dose regimen for each muscle would follow the recommendation of international consensus.
  A. Semitendinosus 5 to 7.5 units/kg of body weight B. Semimembranosus 5 to 7.5 units/kg of body weight C. Gastrocnemius 10 units/kg of body weight D. Maximal total dose per patient : unilateral injection 500 units, bilateral injection 1,000 units E. The dosage of two hamstring muscles will depend on the severity of spasticity and gait abnormalities of children with CP

SUMMARY:
This is a longitudinal, prospective, and open-label interventional study in a single center. We will investigate the effect of single injection in each patient. This study was designed to establish the clinical evidence for effect of botulinum toxin type a (Dysport, abobotulinum toxin A) injection on changes in musculotendinous length and dynamics of hamstring muscles during gait in children with spastic cerebral palsy walking with excessive knee flexion.

Baseline data such as Modified Ashworth scale (MAS), Modified Tardieu scale (MTS), Gross Motor Function Measures (GMFM), and Gross Motor Function Classification System (GMFCS) level will be assessed. Gait analysis will be performed using a computerized gait analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the gait cycle. A trained investigator will place 14 reflective markers on the anterior and posterior superior iliac spine, the mid points of the lateral femur, the lateral knee joint axis, the midpoints of the lateral tibia, the lateral malleolus, and the dorsal foot between metatarsal heads 2 and 3. All subjects should walk barefoot at a self-selected speed along an 8-meter path with the markers in place and the motion will be captured with a 100-Hz sampling frequency. Force-plates (AMTI OR 6-5, Advanced Mechanical Technology, Newton, MA, USA) under the path will record ground reaction forces during the walking trials with a 1000-Hz sampling frequency, and joint moments will be expressed as internal moments to counter the ground reaction forces. Data collection will continue until the subject achieved at least 3 'clean' force-plate strikes. Kinematic and kinetic data from successful trials will be used for statistical analysis. Video recording will be done simultaneously from the front, rear, and side, with the 3D gait analysis.

DETAILED DESCRIPTION:
Based on the evaluation including gait analysis, we will select the target muscles and inject the toxin into the selected muscles of the spastic lower limb under the guidance of ultrasonography or electrical stimulation. After BoNT-A injection, these children will be evaluated after 1 month. Clinical data obtained in the baseline measurement will be assessed again. Motion capture data will also be collected. Finally, clinical data of patients will be collected 4 months after injection to identify the clinical improvement and side effects.

Motion capture data will be imported to OpenSim. We will generate an inverse kinematic analysis of each subject using following procedure:

1. Scale the model to match the anthropometry of each subject. We will scale the dimensions of the torso, pelvis, thigh, shank, and foot based on the relative distances between pairs of markers measured experimentally and the corresponding markers in the model. The muscle attachments will also be scaled with the segment.
2. Using a least-squares formulation, a set of desired joint angles for tracking, consistent with each scaled model, based on the marker trajectories, joint constraints, and joint angles from gait analysis will be computed.
3. The musculotendinous length of each muscle will be calculated based on the "lower limb model 2010" by Arnold. This model adopted the wrapping surface to calculate the moment arm and musculotendinous unit passage at each joint. This model is intended to be used in research-graded kinematic analysis.

   * Objectives <Primary objective>

1.To determine the changes of musculotendinous length of hamstrings after a single BoNT-A injection during walking in children with spastic CP walking with excessive knee flexion <Secondary objectives>

1. To determine the efficacy on gross motor function after BoNT-A injection
2. To determine the benefit on gait after BoNT-A injection
3. To determine the efficacy on spasticity after BoNT-A injection
4. To determine the kinematic change after BoNT-A injection
5. To determine the dynamic change after BoNT-A injection
6. To determine the treatment emergent adverse events following BoNT-A injection

   * Subjects : total 32 children with cerebral palsy
   * Intervention :

1. BoNT-A will be injected into two hamstring and/or gastrocnemius muscles under the guidance of ultrasonography or electrical stimulation. 2. Maximal total dose and dose regimen for each muscle would follow the recommendation of international consensus. A. Semitendinosus 5 to 7.5 units/kg of body weight B. Semimembranosus 5 to 7.5 units/kg of body weight C. Gastrocnemius 10 units/kg of body weight D. Maximal total dose per patient : unilateral injection 500 units, bilateral injection 1,000 units E. The dosage of two hamstring muscles will depend on the severity of spasticity and gait abnormalities of children with CP

* Studies : 3D motion analysis, GMFM (gross motor function measure), GMFCS (gross motor function classification system), MAS (modified Ashworth scale), MTS (modified Tardieu scale)
* Evaluation plan : 1) pre-intervention, 2) post-4 weeks after intervention, 3) 16 weeks after intervention

ELIGIBILITY:
Inclusion Criteria:

* Children with CP over the age of 2 years
* The spasticity is thought to interfere motor learning or cause abnormal posture and movement patterns by "management algorithm" of international consensus.

  1. MAS ≥ 1+ at hamstrings
  2. Dynamic spasticity rather than fixed contracture: Difference between Xv1 and Xv3 is at least 15 degrees in MTS at hamstrings
* I to III levels of GMFCS

Exclusion Criteria:

* Children who received interventions such as chemical nerve block or casting within 6 months
* Children who had baclofen pump
* Children who experienced the adverse reactions from previous BoNT-A injections
* Children who have a mixed type of CP (Athetosis, dystonia) or other movement disorder (eg. ataxia)
* Children who are participating in other investigational study at the moment
* Children who are not suitable for this study according to the investigator's discretion

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-15; Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Changes in musculotendinous length of hamstrings | pre-intervention (1 hour before intervention)
  Changes in musculotendinous length of hamstrings obtained from 3D motion analysis after a single BoNT-A injection during walking in children with spastic CP walking with excessive knee flexion
Changes in musculotendinous length of hamstrings | 4 weeks after intervention
  Changes in musculotendinous length of hamstrings obtained from 3D motion analysis after a single BoNT-A injection during walking in children with spastic CP walking with excessive knee flexion
Changes in musculotendinous length of hamstrings | 16 weeks after intervention
  Changes in musculotendinous length of hamstrings obtained from 3D motion analysis after a single BoNT-A injection during walking in children with spastic CP walking with excessive knee flexion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Severance Hospital, Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No